CLINICAL TRIAL: NCT00298012
Title: Methotrexate in the Treatment of Axial Spondyloarthritis. A Randomized, Multicenter, Double-Blind, Placebo-Controlled Study.
Brief Title: Methotrexate in the Treatment of Axial Spondyloarthritis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Rheumatism Foundation Hospital (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-001202-60
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Spondylarthropathies; Spondylitis, Ankylosing
Keywords: Methotrexate; Magnetic Resonance Imaging; Anterior uveitis
MeSH Terms: conditions — Spondylarthropathies; Spondylitis, Ankylosing; Uveitis, Anterior | interventions — Methotrexate

INTERVENTIONS:
Drug: Methotrexate

SUMMARY:
The goal of this study is to evaluate the efficacy of oral methotrexate for the treatment of active axial spondyloarthritis (early ankylosing spondylitis or spondyloarthritis with sacroiliitis). Efficacy will be measured by reduction in the signs and symptoms of active spondyloarthritis including effects on back pain and stiffness, range of motion in the spine, physical function, quality of life and incidence of arthritis, enthesitis and anterior uveitis.

DETAILED DESCRIPTION:
The established classification criteria for ankylosing spondylitis (AS) rely on the combination of clinical symptoms plus radiographic sacroiliitis of at least grade 2 bilaterally or grade 3 unilaterally. It usually takes several years for definite radiographic sacroiliitis to evolve. Diagnosis of AS may be delayed up to 10 years after the onset of symptoms, if diagnosis is based on the radiographic findings.

A group of leading experts in the field of spondyloarthropathies proposed in 2004 the term "axial spondyloarthritis" as an attempt to narrow the gap of 5-10 years between the first symptoms and the diagnosis of AS (Rudwaleit et al. Ann Rheum Dis 2004; 63:535-43). Using the proposed approach, an early diagnosis of AS (or axial spondyloarthritis) can be made with a high degree of confidence, when at least two to three spondyloarthritis features (clinical findings, laboratory tests or skeletal imaging) are present. Magnetic resonance imaging (MRI) of the sacroiliac joints appears to be especially useful tool in the diagnosis of early AS. Early diagnosis and treatment could probably prevent structural damage and lead to better functional outcomes.

Treatment of AS has largely consisted of non-steroidal anti-inflammatory drugs (NSAIDs). Most disease modifying antirheumatic drugs are not effective in axial manifestations. Sulfasalazine has some efficacy on peripheral symptoms. Tumor necrosis factor (TNF) alpha blocking drugs infliximab and etanercept are effective in both axial and peripheral manifestations of the disease. According to consensus statement, the initiation of anti-TNF alpha therapy requires a definitive diagnosis of AS, which is based on radiographic evidence of sacroiliitis.

It is well documented, that oral methotrexate is effective and safe in the treatment of rheumatoid arthritis and psoriatic arthritis. Still, studies proving its usefulness for the treatment of AS are lacking. To this date, three small randomised and controlled trials to clarify this issue have been conducted. The dose of methotrexate used in these studies was low, only 7,5 - 10 mg per week. One of these studies showed a benefit in the active treatment group. There was no statistically significant benefit of methotrexate in the two other studies.

The purpose of this study is to assess the efficacy of oral methotrexate in adult subjects with active axial spondyloarthritis. Subjects will be randomly assigned to placebo or methotrexate treatment groups. All subjects in the active treatment group receive at least a dose of 15 mg per week of oral methotrexate. To reduce mucosal, gastrointestinal and haematologic side effects of low-dose methotrexate all study subjects receive also a dose of 5 mg per week of folic acid. A stable dose of NSAID during the study is permitted. The duration of the double-blinded treatment period is 24 weeks.

Efficacy of the treatment is measured by reduction in the signs and symptoms of axial spondyloarthritis at weeks 12 and 24. If the primary outcome of ASAS20 (ASsessment in Ankylosing Spondylitis response criteria, improvement of at least 20 % in patient reported symptoms) is not met at the week 12, the dose of methotrexate or corresponding placebo will be increased to 20 mg per week during weeks 12 to 24.

Clinical history of anterior uveitis and its incidence during the study is also recorded. An ophthalmologic examination is performed at baseline and week 24.

To a subset of patients a MRI scan of sacroiliac joints will be done also at week 24, to assess changes of active inflammatory lesions as detected by MRI.

An extension study of radiological progression is also planned. X-ray changes of sacroiliac joints and lumbosacral spine will be assessed at baseline and at 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory back pain (definition in Calin et al. JAMA 1977;237:2613-4) as the presenting symptom,
* Positive laboratory test result for HLA-B27,
* Active sacroiliitis in MRI read by qualified radiologist,
* Active disease despite treatment with at least two NSAIDs.

Active disease is defined as:

1. a score of ≥ 30 mm for morning stiffness (average of 2 scores on a 100 mm visual analog scale [VAS] analysing duration and intensity of morning stiffness),
2. scores of ≥ 30 mm VAS for 2 of the following 3 parameters: patient's global assessment of disease activity, back pain and the Bath Ankylosing Spondylitis Functional Index (BASFI).

Exclusion Criteria:

* Known hypersensitivity to methotrexate
* Have received sulfasalazine within 4 weeks prior to the first administration of study agent
* Using oral corticosteroids on a dose equivalent to ≥10 mg of prednisone/day
* Any concomitant rheumatic disease other than spondyloarthritis
* Fibromyalgia
* Pregnant or breast feeding
* Have had a serious infection within 1 month
* Have any known malignancy or have a history of malignancy within the previous 5 years
* Have current signs or symptoms of severe or uncontrolled renal, hepatic, hematologic, gastrointestinal or pulmonary disease
* Grade 3 or 4 changes in radiographs of sacroiliac joints (grading of radiographs according to the New York criteria)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-03

PRIMARY OUTCOMES:
ASAS20

SECONDARY OUTCOMES:
ASAS40
ASAS5/6
ASAS partial remission
Incidence of arthritis
Incidence of anterior uveitis
BASDAI

CONTACTS AND LOCATIONS:
Overall Officials: Matti Laitinen, MD, Principal Investigator — Rheumatism Foundation Hospital
Locations (5):
- Finland (5):
  - Rheumatism Foundation Hospital, Heinola
  - Helsinki University Central Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere